CLINICAL TRIAL: NCT06918522
Title: Introduction of Sophrology and Art Therapy in Hand and Upper Limb Surgery at Lyon University Hospital
Acronym: ISAT-CCMS
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_1075
Record Dates: First submitted 2025-02-28; First posted 2025-04-09 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Hand and Upper Limb Trauma
Keywords: hand and upper limb trauma; sophrology; art-therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Art-therapy and sophrology evaluation: Each patient eligible for the study will, additionally to the standard care have repeated sessions of sophrology and/or art-therapy along the re-education process. Quality of life as well as anxiety, pain will be assessed before and after each session and at the begining and the end of the re-education process

SUMMARY:
The human and economic impact of hand and upper limb pathologies, whether acute or chronic, surgical or medical, is considerable on a national level. Hand wounds and traumas account for 1/3 of work-related accidents and their consequences. The surgical procedure and its technical quality are essential, but so is the re-education and rehabilitation phase. It is in this post-operative context that sophrology and art therapy could have their place. Literature in this precise field is non-existent. A study is therefore needed to determine the quality of life, feasibility and acceptability of these new techniques in the rehabilitation department of the Édouard Herriot Hospital's Hand and Upper Limb Surgery Unit.

Sophrology and art therapy could help to limit upper-limb sequelae by promoting confidence-building and functional participation, thus helping patients to return more quickly to an active life. Given the current state of knowledge, the hypothesis being tested is that, within the framework of an existing multi-disciplinary team, art therapy and sophrology could improve quality of life and find favorable adherence on the part of patients usually cared for in the upper limb surgery department.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged ≥ 18 years)
* Men and women
* Cared for in the hand and upper limb surgery department as part of emergency or scheduled activity or rehabilitation.
* Wishing to benefit from sophrology and/or art therapy in their care pathway.
* Having expressed his non-opposition

Exclusion Criteria:

* Patients under legal protection
* Any patient who does not have a sufficient command of the language to enable comprehension and expression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized Rehabilitation Department Pavillon T HEH Hospices Civils of Lyon- hand and upper limb surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-22 (Estimated)

PRIMARY OUTCOMES:
Quality of life | Delta between before and after 16 weeks reduction post surgery
  The outcome measure of quality of life will be estimated by the SF12 score (Short-form 12 health survey) in its physical (pain) and mental (anxiety) dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Aram GAZARIAN, Professor, Principal Investigator — Hospices Civils de Lyon. Rehabilitation Department Pavillon T HEH - hand and upper limb surgery
Locations (1):
- Hospices Civils de Lyon. Rehabilitation Department Pavillon T HEH - hand and upper limb surgery, Lyon, France